CLINICAL TRIAL: NCT03629561
Title: Diagnosis of Monoclonal Gammopathy of Renal Significance in Patients With Paraproteinemias
Brief Title: Diagnosis of MGRS in Patients With Paraproteinemias: Clinical, Anatomopathological and Pathophysiological Study
Acronym: MGRS-CAPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academia Nacional de Medicina (Other)
Responsible Party: Principal Investigator, MARIANA CIOCCHINI, Principal Investigator, Academia Nacional de Medicina
Other Study IDs: T.I. N° 12702/18/H
Record Dates: First submitted 2018-08-05; First posted 2018-08-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-07

CONDITIONS: Monoclonal Gammopathy of Renal Significance
Keywords: "Paraproteinemias"[Mesh]; "Kidney Diseases"[Mesh]

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood,Urine,Renal tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is the first prospective study which evaluate patients with small B-cell clones to diagnose monoclonal gammopathy of renal significance (MGRS) and characterize it clinically, anatomopathologically and pathophysiologically taking int account a geriatric approach.

ELIGIBILITY:
Inclusion Criteria:

* Paraproteinemias

Exclusion Criteria:

* Multiple Myeloma
* Waldenstrom Macroglobulinemia
* Chronic Lymphocytic Leukemia
* Malignant Lymphoma
* Monoclonal gammopathy of unknown significance (MGUS) secondary to Infections
* MGUS secondary to Autoimmune Diseases
* Uncompleted hematological evaluation
* Renal tumor except for cysts Bosniak type I/II
* Other malignant neoplasia
* Unresolved obstructive uropathy
* Patients with only one kidney except for renal transplant
* Co-morbidities which would limit the ability to receive aggressive therapeutic intervention
* Fragile old people
* Pregnancy
* Prison
* Impatient in psychiatric institutions.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematological or nephrological patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-02-23 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Renal histopathology compatible with MGRS | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Renal physiopathological changes | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Academia Nacional de Medicina, Buenos Aires, Argentina

REFERENCES:
- [Background] Ciocchini M, Arbelbide J, Musso CG. Monoclonal gammopathy of renal significance (MGRS): the characteristics and significance of a new meta-entity. Int Urol Nephrol. 2017 Dec;49(12):2171-2175. doi: 10.1007/s11255-017-1594-y. Epub 2017 Apr 19. PMID 28425076
- [Background] Ciocchini M, Musso CG. What is the place of POEMS syndrome in the current classification of monoclonal gammopathies of renal significance? Int Urol Nephrol. 2018 Feb;50(2):383-384. doi: 10.1007/s11255-017-1739-z. Epub 2017 Nov 13. No abstract available. PMID 29134615
- [Background] Ciocchini M, Musso CG. Which should be the correct treatment for monoclonal gammopathy of renal significance with complement alternative pathway dysregulation (C3 glomerulopathy and atypical hemolytic uremic syndrome): clone-directed or anticomplement therapy? Int Urol Nephrol. 2018 Jul;50(7):1365-1366. doi: 10.1007/s11255-018-1896-8. Epub 2018 May 28. No abstract available. PMID 29808447
- [Background] Rosner MH, Edeani A, Yanagita M, Glezerman IG, Leung N; American Society of Nephrology Onco-Nephrology Forum. Paraprotein-Related Kidney Disease: Diagnosing and Treating Monoclonal Gammopathy of Renal Significance. Clin J Am Soc Nephrol. 2016 Dec 7;11(12):2280-2287. doi: 10.2215/CJN.02920316. Epub 2016 Aug 15. PMID 27526705
- [Background] Chauvet S, Fremeaux-Bacchi V, Petitprez F, Karras A, Daniel L, Burtey S, Choukroun G, Delmas Y, Guerrot D, Francois A, Le Quintrec M, Javaugue V, Ribes D, Vrigneaud L, Arnulf B, Goujon JM, Ronco P, Touchard G, Bridoux F. Treatment of B-cell disorder improves renal outcome of patients with monoclonal gammopathy-associated C3 glomerulopathy. Blood. 2017 Mar 16;129(11):1437-1447. doi: 10.1182/blood-2016-08-737163. Epub 2017 Jan 9. PMID 28069603
- [Background] Leung N, Nasr SH. A Patient with Abnormal Kidney Function and a Monoclonal Light Chain in the Urine. Clin J Am Soc Nephrol. 2016 Jun 6;11(6):1073-1082. doi: 10.2215/CJN.10641015. Epub 2016 Mar 18. PMID 26992418
- [Background] Motwani SS, Herlitz L, Monga D, Jhaveri KD, Lam AQ; American Society of Nephrology Onco-Nephrology Forum. Paraprotein-Related Kidney Disease: Glomerular Diseases Associated with Paraproteinemias. Clin J Am Soc Nephrol. 2016 Dec 7;11(12):2260-2272. doi: 10.2215/CJN.02980316. Epub 2016 Aug 15. PMID 27526706
- [Background] Fish R, Pinney J, Jain P, Addison C, Jones C, Jayawardene S, Booth J, Howie AJ, Ghonemy T, Rajabali S, Roberts D, White L, Khan S, Morgan M, Cockwell P, Hutchison CA. The incidence of major hemorrhagic complications after renal biopsies in patients with monoclonal gammopathies. Clin J Am Soc Nephrol. 2010 Nov;5(11):1977-80. doi: 10.2215/CJN.00650110. Epub 2010 Jul 22. PMID 20651154
- [Background] Sethi S, D'Agati VD, Nast CC, Fogo AB, De Vriese AS, Markowitz GS, Glassock RJ, Fervenza FC, Seshan SV, Rule A, Racusen LC, Radhakrishnan J, Winearls CG, Appel GB, Bajema IM, Chang A, Colvin RB, Cook HT, Hariharan S, Herrera Hernandez LP, Kambham N, Mengel M, Nath KA, Rennke HG, Ronco P, Rovin BH, Haas M. A proposal for standardized grading of chronic changes in native kidney biopsy specimens. Kidney Int. 2017 Apr;91(4):787-789. doi: 10.1016/j.kint.2017.01.002. PMID 28314581
- [Background] Moutzouris DA, Herlitz L, Appel GB, Markowitz GS, Freudenthal B, Radhakrishnan J, D'Agati VD. Renal biopsy in the very elderly. Clin J Am Soc Nephrol. 2009 Jun;4(6):1073-82. doi: 10.2215/CJN.00990209. Epub 2009 May 14. PMID 19443626
- [Background] Trimarchi H, Barratt J, Cattran DC, Cook HT, Coppo R, Haas M, Liu ZH, Roberts IS, Yuzawa Y, Zhang H, Feehally J; IgAN Classification Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Conference Participants. Oxford Classification of IgA nephropathy 2016: an update from the IgA Nephropathy Classification Working Group. Kidney Int. 2017 May;91(5):1014-1021. doi: 10.1016/j.kint.2017.02.003. Epub 2017 Mar 22. PMID 28341274
- [Background] Javaugue V, Bouteau I, Sirac C, Quellard N, Diolez J, Colombo A, Desport E, Ecotiere L, Goujon JM, Fermand JP, Touchard G, Jaccard A, Bridoux F. [Classification and therapeutic management of monoclonal gammopathies of renal significance]. Rev Med Interne. 2018 Mar;39(3):161-170. doi: 10.1016/j.revmed.2017.03.012. Epub 2017 Apr 27. French. PMID 28457684
- [Background] Borza DB, Chedid MF, Colon S, Lager DJ, Leung N, Fervenza FC. Recurrent Goodpasture's disease secondary to a monoclonal IgA1-kappa antibody autoreactive with the alpha1/alpha2 chains of type IV collagen. Am J Kidney Dis. 2005 Feb;45(2):397-406. doi: 10.1053/j.ajkd.2004.09.029. PMID 15685519
- [Background] Vignon M, Cohen C, Faguer S, Noel LH, Guilbeau C, Rabant M, Higgins S, Hummel A, Hertig A, Francois H, Lequintrec M, Vilaine E, Knebelmann B, Pourrat J, Chauveau D, Goujon JM, Javaugue V, Touchard G, El Karoui K, Bridoux F. The clinicopathologic characteristics of kidney diseases related to monotypic IgA deposits. Kidney Int. 2017 Mar;91(3):720-728. doi: 10.1016/j.kint.2016.10.026. Epub 2017 Jan 6. PMID 28069266
- [Background] Stokes MB, Valeri AM, Herlitz L, Khan AM, Siegel DS, Markowitz GS, D'Agati VD. Light Chain Proximal Tubulopathy: Clinical and Pathologic Characteristics in the Modern Treatment Era. J Am Soc Nephrol. 2016 May;27(5):1555-65. doi: 10.1681/ASN.2015020185. Epub 2015 Sep 15. PMID 26374607
- [Background] Eirin A, Irazabal MV, Gertz MA, Dispenzieri A, Lacy MQ, Kumar S, Sethi S, Nasr SH, Cornell LD, Fidler ME, Fervenza FC, Leung N. Clinical features of patients with immunoglobulin light chain amyloidosis (AL) with vascular-limited deposition in the kidney. Nephrol Dial Transplant. 2012 Mar;27(3):1097-101. doi: 10.1093/ndt/gfr381. Epub 2011 Nov 7. PMID 22067518
- [Background] Sicard A, Karras A, Goujon JM, Sirac C, Bender S, Labatut D, Callard P, Sarkozy C, Essig M, Vanhille P, Provot F, Nony A, Nochy D, Ronco P, Bridoux F, Touchard G. Light chain deposition disease without glomerular proteinuria: a diagnostic challenge for the nephrologist. Nephrol Dial Transplant. 2014 Oct;29(10):1894-902. doi: 10.1093/ndt/gfu045. Epub 2014 Mar 11. PMID 24619059
- [Background] Messias NC, Walker PD, Larsen CP. Paraffin immunofluorescence in the renal pathology laboratory: more than a salvage technique. Mod Pathol. 2015 Jun;28(6):854-60. doi: 10.1038/modpathol.2015.1. Epub 2015 Feb 13. PMID 25676556
- [Background] Larsen CP, Ambuzs JM, Bonsib SM, Boils CL, Cossey LN, Messias NC, Silva FG, Wang YH, Gokden N, Walker PD. Membranous-like glomerulopathy with masked IgG kappa deposits. Kidney Int. 2014 Jul;86(1):154-61. doi: 10.1038/ki.2013.548. Epub 2014 Jan 15. PMID 24429395
- [Background] Ramirez-Alvarado M, Barnidge DR, Murray DL, Dispenzieri A, Marin-Argany M, Dick CJ, Cooper SA, Nasr SH, Ward CJ, Dasari S, Jimenez-Zepeda VH, Leung N. Assessment of renal response with urinary exosomes in patients with AL amyloidosis: A proof of concept. Am J Hematol. 2017 Jun;92(6):536-541. doi: 10.1002/ajh.24717. Epub 2017 May 4. PMID 28295502
- [Background] Sharma SG, Bomback AS, Radhakrishnan J, Herlitz LC, Stokes MB, Markowitz GS, D'Agati VD. The modern spectrum of renal biopsy findings in patients with diabetes. Clin J Am Soc Nephrol. 2013 Oct;8(10):1718-24. doi: 10.2215/CJN.02510213. Epub 2013 Jul 25. PMID 23886566
- [Background] Paueksakon P, Revelo MP, Horn RG, Shappell S, Fogo AB. Monoclonal gammopathy: significance and possible causality in renal disease. Am J Kidney Dis. 2003 Jul;42(1):87-95. doi: 10.1016/s0272-6386(03)00412-8. PMID 12830460
- [Background] Hutchison CA, Harding S, Hewins P, Mead GP, Townsend J, Bradwell AR, Cockwell P. Quantitative assessment of serum and urinary polyclonal free light chains in patients with chronic kidney disease. Clin J Am Soc Nephrol. 2008 Nov;3(6):1684-90. doi: 10.2215/CJN.02290508. PMID 18945993
- [Background] Helal I, Fick-Brosnahan GM, Reed-Gitomer B, Schrier RW. Glomerular hyperfiltration: definitions, mechanisms and clinical implications. Nat Rev Nephrol. 2012 Feb 21;8(5):293-300. doi: 10.1038/nrneph.2012.19. PMID 22349487
- [Background] Cachat F, Combescure C, Cauderay M, Girardin E, Chehade H. A systematic review of glomerular hyperfiltration assessment and definition in the medical literature. Clin J Am Soc Nephrol. 2015 Mar 6;10(3):382-9. doi: 10.2215/CJN.03080314. Epub 2015 Jan 7. PMID 25568216
- [Background] Schaeffner ES, Ebert N, Delanaye P, Frei U, Gaedeke J, Jakob O, Kuhlmann MK, Schuchardt M, Tolle M, Ziebig R, van der Giet M, Martus P. Two novel equations to estimate kidney function in persons aged 70 years or older. Ann Intern Med. 2012 Oct 2;157(7):471-81. doi: 10.7326/0003-4819-157-7-201210020-00003. PMID 23027318
- [Background] Saeki T, Kawano M. IgG4-related kidney disease. Kidney Int. 2014 Feb;85(2):251-7. doi: 10.1038/ki.2013.393. Epub 2013 Oct 9. PMID 24107849
- [Background] Musso CG, Reynaldi J, Martinez B, Pierangelo A, Vilas M, Algranati L. Renal reserve in the oldest old. Int Urol Nephrol. 2011 Mar;43(1):253-6. doi: 10.1007/s11255-010-9769-9. Epub 2010 Jul 1. PMID 20593305
- [Background] Jhaveri KD, Shah HH, Patel C, Kadiyala A, Stokes MB, Radhakrishnan J. Glomerular diseases associated with cancer, chemotherapy, and hematopoietic stem cell transplantation. Adv Chronic Kidney Dis. 2014 Jan;21(1):48-55. doi: 10.1053/j.ackd.2013.08.003. PMID 24359986